CLINICAL TRIAL: NCT06498674
Title: Clinical Application of AI-assisted Ultrasound Technology in the Preoperative Evaluation of Thyroid Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor Affiliation: Fujian Medical University Collaborators:, Fujian Medical University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AI-base PCD
Record Dates: First submitted 2024-06-09; First posted 2024-07-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; Artificial Intelligence; Ultrasound; Preoperative Assessment
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concordant Group (Other): Patients in whom the detection and diagnostic results of thyroid nodules and lymph nodes are consistent between traditional two-dimensional ultrasound and AI-assisted ultrasound.
  Interventions: Other: No Need for Supplementary Pathological Examination
- Discordant Group (Other): Patients in whom the detection and diagnostic results of thyroid nodules and lymph nodes differ between traditional two-dimensional ultrasound and AI-assisted ultrasound.
  Interventions: Diagnostic Test: Supplementary Pathological Examination

INTERVENTIONS:
Diagnostic Test: Supplementary Pathological Examination — For the same thyroid nodule, if there is discordance between the interpretations of AI-assisted ultrasound and traditional two-dimensional ultrasound, supplementary fine needle aspiration biopsy or intraoperative biopsy will be performed to clarify the nature of the nodule.
  Arms: Discordant Group
Other: No Need for Supplementary Pathological Examination — For the same thyroid nodule, if there is discordance between the interpretations of AI-assisted ultrasound and traditional two-dimensional ultrasound, there is no need for supplementary fine needle aspiration biopsy or intraoperative biopsy.
  Arms: Concordant Group

SUMMARY:
This study aims to explore the application of AI-assisted ultrasound technology in the preoperative assessment of thyroid cancer. Traditional ultrasound examination data from thyroid cancer patients will be collected, and AI systems will be utilized to detect and diagnose thyroid nodules and lymph nodes. In cases where there is disagreement between the two-dimensional ultrasound and AI system results, further confirmation will be sought through biopsy. Subsequently, pathological results will serve as the "gold standard" for comparison between the AI system and traditional ultrasound examination results, assessing their accuracy and reliability. Through this research endeavor, a more accurate and reliable method for preoperative assessment of thyroid cancer is aspired to be offered, thereby supporting clinical decision-making and paving the way for novel applications of AI in the field of medical imaging diagnosis.

DETAILED DESCRIPTION:
This study aims to investigate the application of AI-assisted ultrasound technology in the preoperative assessment of thyroid cancer. Traditional ultrasound examination data from patients with thyroid cancer, including two-dimensional ultrasound images, color Doppler flow images, and detailed characteristics of thyroid nodules and lymph nodes such as number, size, morphology, echogenicity, margins, calcifications, and aspect ratio, will be collected. Prior to surgery, a reassessment will be conducted using AI-assisted ultrasound technology, and the detection and diagnostic results of thyroid nodules and lymph nodes by the AI system will be recorded. In cases where there is discrepancy between the results of two-dimensional ultrasound and the AI system, fine needle aspiration biopsy or intraoperative biopsy will be performed for further confirmation of their nature. Post-surgery, the pathological results of each nodule will serve as the "gold standard" for comparative analysis between the AI system and traditional two-dimensional ultrasound examinations. The accuracy of the AI system in detecting and localizing nodules will be analyzed, and its sensitivity, specificity, and accuracy will be calculated to evaluate its diagnostic efficacy and reliability in the preoperative assessment of thyroid cancer. Through this research, a more accurate and reliable adjunctive diagnostic method for the preoperative assessment of thyroid cancer is aimed to be provided to assist clinical decision-making. Additionally, new avenues and directions for the application of AI in the field of medical imaging diagnosis will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preoperative pathological confirmation of thyroid malignant tumors undergoing surgical treatment.
* Patients with benign thyroid tumors, such as thyroid adenomas causing compressive symptoms, undergoing surgical treatment.
* Patients with complete and high-quality traditional two-dimensional color ultrasound images.
* Complete postoperative pathology reports.
* Willingness to participate in this clinical trial and signing of informed consent.

Exclusion Criteria:

* Patients with a history of neck surgery or radiotherapy.
* Patients with a history of malignant tumors in other parts of the body.
* Patients with thyroid dysfunction.
* Incomplete or poor-quality traditional two-dimensional color ultrasound images.
* Incomplete postoperative pathology reports.
* Refusal to participate in this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Supplementary Pathological Examination | One day after surgery
  For patients who have completed traditional two-dimensional color ultrasound and AI-assisted ultrasound, record whether a supplementary pathological examination was conducted.
Change in Treatment Decision | One day after surgery
  For patients who have completed traditional two-dimensional color ultrasound, AI-assisted ultrasound, and undergone supplementary pathological examination, record whether there was a change in the surgical approach or scope.

SECONDARY OUTCOMES:
Traditional Two-Dimensional Color Ultrasound Findings | Preoperative
  Record ultrasound image features such as number, size, morphology, echogenicity, margins, calcifications, and TI-RADS score of thyroid nodules and lymph nodes under traditional two-dimensional color ultrasound.
AI-Assisted Ultrasound Interpretation Results | Preoperative
  Record ultrasound image features such as number, size, morphology, echogenicity, margins, calcifications, and TI-RADS score of thyroid nodules and lymph nodes under AI-assisted ultrasound.
Supplementary Pathological Examination Results | One day Postoperative
  For patients who underwent supplementary pathological examination, record the results of their pathological examination.
Postoperative Pathology Report | One day after the postoperative pathology report is released
  Record the presence of thyroid lesions and lymph node metastasis in the postoperative pathology report.
Statistical Indicators | One day after the postoperative pathology report is released
  Using pathological evidence as the gold standard, construct contingency tables for both preoperative traditional two-dimensional color ultrasound and AI-assisted ultrasound, calculate sensitivity, specificity
Statistical Indicator missed diagnosis rate. | One day after the postoperative pathology report is released
  Using pathological evidence as the gold standard, construct contingency tables for both preoperative traditional two-dimensional color ultrasound and AI-assisted ultrasound, missed diagnosis rate.
Statistical Indicator positive predictive value | One day after the postoperative pathology report is released
  Using pathological evidence as the gold standard positive predictive value
Statistical Indicator Youden index | One day after the postoperative pathology report is released
  Using pathological evidence as the gold standard Youden index.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China